CLINICAL TRIAL: NCT05340439
Title: Prospective, Open-label, Non-randomized, Single-arm, Dose Titration Study to Investigate the Efficacy and Safety of IncobotulinumtoxinA in Children Deemed to Require a Total Body Dose up to 22U/kg (Maximum Dose 550U) During the Study Period for the Treatment of Upper and Lower Limb Spasticity Due to Cerebral Palsy
Brief Title: INcobotulinumtoxina in ChIldren Upper and Lower Limb sPasticITy (INCIPIT)
Acronym: INCIPIT
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Responsible Party: Principal Investigator, Nicola Smania, MD, Clinical Professor, Prof., Universita di Verona
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: INCIPIT
Record Dates: First submitted 2022-04-07; First posted 2022-04-22 (Actual); Last update posted 2022-04-22 (Actual); Status verified 2022-04

CONDITIONS: Spastic Cerebral Palsy
Keywords: Cerebral Palsy; Botulinum toxin type A; Spasticity; Titration study
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — incobotulinumtoxinA

STUDY DESIGN:
Intervention Model Description: Prospective, open-label, non-randomized, single-arm, dose titration, phase II study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Incobotulinumtoxin A treatment (Experimental): The study will consist of three injection cycles. In each, an injection visit is followed by an observation period of 12 to 20 weeks.
  Interventions: Drug: IncobotulinumtoxinA 100 UNT [Xeomin]

INTERVENTIONS:
Drug: IncobotulinumtoxinA 100 UNT [Xeomin] — In cycle 1, a total body dose of 16U/kg (maximum 400U) of IncobotulinumtoxinA will be injected into the spastic muscles of the affected limbs.
  In cycle 2, a total body dose of 19U/kg (maximum 475U) of IncobotulinumtoxinA will be injected. If a dose of 19U/kg is not justified (i.e., for clinical or safety reasons) but BoNT-A treatment is still needed (according to the clinical condition of patients) the same dose injected in cycle 1 (16U/Kg; maximum 400U) may be administered in the cycle 2.
  In cycle 3, a total body dose of 22U/kg (maximum 550U) of IncobotulinumtoxinA will be injected. If a dose of 22U/kg is not justified (i.e., for clinical or safety reasons) but BoNT-A treatment is still needed (according to the clinical condition of patients) the same dose injected in cycle 2 (19U/Kg; maximum 600U) may be administered in the cycle 3 (if the patient has been treated with 16U/kg in cycle 2, a dose of 19U/kg may be injected in cycle 3).

SUMMARY:
Prospective, open-label, non-randomized, single-arm, dose titration, phase II study.

The study will consist of three injection cycles. In each, an injection visit is followed by an observation period of 12 to 20 weeks.

During cycle 1, a total body dose of 16U/kg (maximum 400U) of IncobotulinumtoxinA will be injected into the spastic muscles of the affected limbs.

During cycle 2, a total body dose of 19U/kg (maximum 475U) of IncobotulinumtoxinA will be injected into the spastic muscles of the affected limbs. If a dose of 19U/kg is not justified (i.e., for clinical or safety reasons) but BoNT-A treatment is still needed (according to the clinical condition of patients) the same dose injected in cycle 1 (16U/Kg; maximum 400U) may be administered in the cycle 2.

During cycle 3, a total body dose of 22U/kg (maximum 550U) of IncobotulinumtoxinA will be injected into the spastic muscles of the affected limbs. If a dose of 22U/kg is not justified (i.e., for clinical or safety reasons) but BoNT-A treatment is still needed (according to the clinical condition of patients) the same dose injected in cycle 2 (19U/Kg; maximum 475U) may be administered in the cycle 3.

DETAILED DESCRIPTION:
The population involved will be children (either BoNT-A treatment-naïve or pre-treated) with multifocal spasticity of the upper and lower limb due to cerebral palsy, scheduled to receive at least one dose of 16 U/kg (maximum 400U) of IncobotulinumtoxinA. No stratification by gender or age is planned.

Our main aim will be to investigate the efficacy of IncobotulinumtoxinA in the treatment of both BoNT-A naïve and pretreated children for upper and lower limb spasticity using a dose titration approach over three injection cycles, with a flexible observation period after injection of 12 to 20 weeks and a total duration of exposure up to 60 weeks.

Our secondary aim will be to investigate the safety of IncobotulinumtoxinA in the treatment of both BoNT-A naïve and pretreated children for upper and lower limb spasticity using a dose titration approach over three injection cycles, with a flexible observation period after injection of 12 to 20 weeks and a total duration of exposure up to 60 weeks.

Treatment procedures BoNT-A has been established as effective and safe (Level A recommendation) for the treatment of childhood spasticity in CP [18]. It acts in the cytosol of nerve endings and inhibits the release of acetylcholine at neuromuscular junctions by cleaving the synaptosomal-associated protein of 25kDa, which is required for vesicle docking and, consequently, neurotransmitter release. BoNT-A injections guided by ultrasonography are allowed into the spastic muscle affected limbs of both body sides.

Considering a dose of 16 U/kg (maximum 400U) licensed for OnabotulinumoxinA and a conversion ratio of 1:1 between OnabotulinumtoxinA and IncobotulinumtoxinA was defined the following dose for cycle 1 according to Law 648/96. Dose titration was defined according to the previous evidence in adults coming from the Tower study [10].

In cycle 1, a total body dose of 16U/kg (maximum 400U) of IncobotulinumtoxinA will be injected into the spastic muscles of the affected limbs.

In cycle 2, a total body dose of 19U/kg (maximum 475U) of IncobotulinumtoxinA will be injected into the spastic muscles of the affected limbs. If a dose of 19U/kg is not justified (i.e., for clinical or safety reasons) but BoNT-A treatment is still needed (according to the clinical condition of patients) the same dose injected in cycle 1 (16U/Kg; maximum 400U) may be administered in the cycle 2.

In cycle 3, a total body dose of 22U/kg (maximum 550U) of IncobotulinumtoxinA will be injected into the spastic muscles of the affected limbs. If a dose of 22U/kg is not justified (i.e., for clinical or safety reasons) but BoNT-A treatment is still needed (according to the clinical condition of patients) the same dose injected in cycle 2 (19U/Kg; maximum 600U) may be administered in the cycle 3 (if the patient has been treated with 16U/kg in cycle 2, a dose of 19U/kg may be injected in cycle 3).

As to cycles 2 and 3, the following clinical and safety issues will be considered to not justify the dose increase to 19U/kg or 22U/kg: full achievement of the goals set on the GAS as a consequence of a clinically significant reduction of treated muscle tone (quantifiable in at least 1 point on the AS); occurrence of the adverse events reported in paragraph 7 (risks and benefits) and not included in the "withdrawal criteria".

Concomitant therapies

Co-administration of the following drugs will not be allowed during the study period:

* Aminoglycoside antibiotics
* Spectinomycin
* Agents interfering with neuromuscular transmission (e.g. tubocurarine-type muscle relaxants)
* 4-Aminoquinoline
* Anticholinergic drugs
* AbobotulinumtoxinA (Dysport) and OnabotulinumtoxinA (Botox) Thus, in case these drugs will be needed/administered, the patient will have to withdraw from the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with upper and lower limb spasticity due to cerebral palsy
* Gross Motor Function Classification System (GMFCS) from Level II to Level V
* Selected target clinical pattern diagnosed by a qualified health care professional (i.e. physiatrist)
* Focal spasticity scored at least 2 points on the Ashworth scale (AS) in the joints associated with the selected target clinical pattern
* Patient deemed by the investigator to require a total body dose up to 22U/kg (maximum 550U) during the study period
* In the case of children pretreated with BoNT-A, time from the last injection at least 5 months
* Informed consent signed by parents or legal guardian.

Exclusion Criteria:

* Participation in other trials
* BoNT-A treatment contraindicated
* Therapy with anticoagulants or other substances that could have an anticoagulant effect
* Girls of childbearing potential (defined as females post menarche)
* Presence of fixed contractures, or bony deformities of the affected limbs
* Previous treatment of spastic muscles with nerve penalization
* Other neurological or orthopaedic conditions involving the affected limbs.

Specific vulnerable populations:

* institutionalized patients will not be included
* girls of childbearing potential (defined as females with a history of menarche) will not be included.

Withdrawal criteria for single patients:

* Serious adverse event (SAE)
* Development of dysphagia and/or aspiration pneumonia.
* Withdrawal of consent
* Inability to follow the study according to its design and time points
* Co-administration of aminoglycoside antibiotics, spectinomycin, 4-aminoquinoline, anticholinergic drugs, AbobotulinumtoxinA, OnabotulinumtoxinA or other agents interfering with neuromuscular transmission (e.g., tubocurarine-type muscle relaxants).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2024-01 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
Ashworth Scale | During the screening assessment
  The Ashworth scale is a well-known and commonly used scale in clinical trials with spasticity. It will be used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Ashworth Scale | Immediately before each IncobotulinumtoxinA treatment session
  The Ashworth scale is a well-known and commonly used scale in clinical trials with spasticity. It will be used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Ashworth Scale | During the follow-up clinical assessment at 4 weeks from each injection
  The Ashworth scale is a well-known and commonly used scale in clinical trials with spasticity. It will be used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).
Ashworth Scale | During the follow-up clinical assessment at 12 weeks from each injection
  The Ashworth scale is a well-known and commonly used scale in clinical trials with spasticity. It will be used to categorize the severity of spasticity by judging resistance to passive movement. It is a 5-point scale that ranges from 0 (=no increase in tone) to 4 (=limb rigid in flexion or extension).

SECONDARY OUTCOMES:
REsistance to PAssive movement Scale (REPAS) | Immediately before each IncobotulinumtoxinA treatment session; at the follow-up clinical assessment at 4 and 12 weeks from each injection
  The REPAS is a summary 26-item test used to assess resistance to passive movement in all four limbs of the body. It provides a global evaluation of spasticity status, as well as per hemibody and per limb. 16 items describe the condition of both upper limbs, 10 that of both lower limbs. Each item is rated by using the AS. The sum of the values represent the REPAS score which may range from zero (no resistance for any item) to 104 (limbs rigid for all items).
Gross Motor Function Classification System (GMFCS) | During the screening assessment; immediately before each IncobotulinumtoxinA treatment session; at the follow-up clinical assessment at 4 and 12 weeks from each injection
  Is a 5 level classification system that describes the gross motor function of people with cerebral palsy (I=can walk indoors and outdoors and climb stairs without using hands for support; II=can climb stairs with a railing, has difficulty with uneven surfaces, inclines or in crowds; III=walks with assistive mobility devices indoors and outdoors on level surfaces, may be able to climb stairs using a railing, may propel a manual wheelchair and need assistance for long distances or uneven surfaces; IV=walking ability severely limited even with assistive devices, uses wheelchairs most of the time and may propel own power wheelchair, standing transfers, with or without assistance; V=has physical impairments that restrict voluntary control of movement, ability to maintain head and neck position against gravity restricted, impaired in all areas of motor function, cannot sit or stand independently, even with adaptive equipment).
Visual Analog Scale (VAS) | Immediately before each IncobotulinumtoxinA treatment session; at the follow-up clinical assessment at 4 and 12 weeks from each injection
  The VAS, which is a validated, subjective measure for acute and chronic pain. Scores are recorded by making a handwritten mark on a 10-cm line that represents a continuum between "no pain" and "worst pain."
Goal Attainment scale (GAS) | Immediately before each IncobotulinumtoxinA treatment session; at the follow-up clinical assessment at 4 and 12 weeks from each injection
  The GAS measures the extent to which a subject's individual goals are achieved in course of intervention. The subject and treating team have to identify 2 personal goals for each treated limb at each injection cycle. Investigator rates the GAS score for each injection cycle. The degree of goal attainment is rated on a 5-point scale (-2, -1, 0, +1, +2; study baseline set to -1) and in order to account for interindividual differences in the number of goals (positive values indicate higher goal attainment).
Global Assessment of Efficacy | At the follow-up clinical assessment at 4 and 12 weeks from each injection
  The Global Assessment of Efficacy, which will be assessed by the investigator, the patient (if possible), and the caregiver using a 4-point Likert scale with the ratings 1 = very good, 2 =good, 3 = moderate, and 4 = poor.
Global Assessment of Tolerability | At the follow-up clinical assessment at 4 and 12 weeks from each injection
  The Global Assessment of Tolerability, which will be assessed by the investigator at each injection cycle control [V3, V6, V9] and end of cycle visits [V4, V7, V10] using a 4-point Likert scale with the ratings 1 = very good, 2 = good, 3 = moderate, and 4 = poor.

IPD SHARING:
Plan to Share IPD: No